CLINICAL TRIAL: NCT05355818
Title: A Phase 3 Clinical Trial to Evaluate Efficacy and Safety of Twice-daily Applications of Delgocitinib Cream 20 mg/g Compared With Cream Vehicle for a 16-week Treatment Period in Adolescents 12-17 Years of Age With Moderate to Severe Chronic Hand Eczema (DELTA TEEN)
Brief Title: Efficacy and Safety of Delgocitinib Cream in Adolescents 12-17 Years of Age With Moderate to Severe Chronic Hand Eczema
Acronym: DELTA TEEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LP0133-1426; 2021-006340-27 (EudraCT Number); U1111-1284-2122 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hand Eczema
MeSH Terms: interventions — delgocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delgocitinib cream (Experimental): Delgocitinib cream 20 mg/g twice daily
  Interventions: Drug: Delgocitinib
- Cream vehicle (Placebo Comparator): Cream vehicle twice daily
  Interventions: Drug: Cream vehicle

INTERVENTIONS:
Drug: Delgocitinib — Cream for topical application
  Arms: Delgocitinib cream
Drug: Cream vehicle — The cream vehicle is similar to the delgocitinib cream except that it does not contain any active medical ingredient.
  Arms: Cream vehicle

SUMMARY:
The purpose of this trial is to test if delgocitinib cream is effective in treating chronic hand eczema (CHE) and to find out what side effects it may have compared with a cream vehicle with no active medical ingredient in adolescents aged 12-17 years. At each visit to the clinic, the doctor will assess the severity and extent of CHE, and during the trial, the adolescents will assess their CHE signs and symptoms as well as quality of life.

The trial will last up to 22 weeks and has a 1-4 week screening period, a 16-week treatment period and a 2- week follow-up period. During the treatment period, each adolescent participant will use either the delgocitinib cream or cream vehicle twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 17 years at screening and baseline.
* Diagnosis of CHE, defined as hand eczema that has persisted for more than 3 months or returned twice or more within the last 12 months.
* Disease severity graded as moderate to severe at screening and baseline according to IGA CHE (i.e. an IGA-CHE score of 3 or 4).
* Subjects who have a documented recent history of inadequate response to treatment with topical corticosteroids (TCS) (at any time within 1 year before the screening visit) or for whom TCS are documented to be otherwise medically inadvisable (e.g. due to important side effects or safety risks).

  * Inadequate response is defined as a history of failure to achieve and maintain a low disease activity state (comparable to an IGA-CHE score of ≤2) despite treatment with a daily regimen of TCS of class III-IV (potent to very potent) for Europe and Australia and class IV-I (medium potency to very/ultra-high potency) for Canada, applied for at least 28 days or for the maximum duration recommended by the product prescribing information, whichever is shorter.
  * Important side effects or safety risks are those that outweigh the potential treatment benefits and include intolerance to treatment, hypersensitivity reactions, and significant skin atrophy as assessed by the physician.

Exclusion Criteria:

* Concurrent skin diseases on the hands, e.g. tinea manuum.
* Clinically significant infection (e.g. impetiginised hand eczema) on the hands.
* Systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine), immunomodulating drugs, retinoids (e.g. alitretinoin), or corticosteroids within 28 days prior to baseline (steroid eyedrops and inhaled or intranasal steroids corresponding to up to 1 mg prednisolone for allergic conjunctivitis, asthma, or rhinitis are allowed).
* Use of tanning beds, phototherapy (e.g. ultraviolet B (UVB), ultraviolet A1 (UVA1), psoralen ultraviolet A (PUVA)), or bleach baths on the hands within 28 days prior to baseline.
* Previous or current treatment with JAK inhibitors (including delgocitinib/LEO 124249), systemic or topical.
* Cutaneously applied treatment with immunomodulators (e.g. PDE-4 inhibitors, pimecrolimus, tacrolimus) or TCS on the hands within 14 days prior to baseline.
* Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 14 days prior to baseline.
* Other cutaneously applied therapy on the hands (except for the use of subject's own emollients) within 7 days prior to baseline.
* Cutaneously applied treatments in regions other than the hands, which could interfere with clinical trial evaluations or pose a safety concern within 7 days prior to baseline.
* Any disorder which is not stable and could:

  * Affect the safety of the subject throughout the trial.
  * Impede the subject's ability to complete the trial. Examples include but are not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, immunological, and psychiatric disorders, and major physical impairment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (35):
- Australia (4):
  - LEO Pharma investigational site, Darlinghurst
  - LEO Pharma investigational site, Mitcham
  - LEO Pharma investigational site, Phillip
  - LEO Pharma investigational site, Woolloongabba
- Belgium (4):
  - LEO Pharma investigational site, Brussels
  - LEO Pharma investigational site, Ghent
  - LEO Pharma investigational site, Gilly
  - LEO Pharma investigational site, Liège
- Canada (8):
  - LEO Pharma investigational site, Edmonton
  - LEO Pharma investigational site, Fredericton
  - LEO Pharma investigational site, Kingston
  - LEO Pharma investigational site, Montreal
  - LEO Pharma investigational site, Red Deer
  - LEO Pharma investigational site, St. John's
  - LEO Pharma investigational site, Toronto
  - LEO Pharma investigational site, Winnipeg
- France (4):
  - LEO Pharma investigational site, Martigues, Bouches-du-Rhône
  - LEO Pharma investigational site, Nice
  - LEO Pharma investigational site, Reims
  - LEO Pharma investigational site, Toulouse
- Poland (4):
  - LEO Pharma investigational site, Chorzów
  - LEO Pharma investigational site, Krakow
  - LEO Pharma investigational site, Warsaw
  - LEO Pharma investigational site, Wroclaw
- Spain (6):
  - LEO Pharma investigational site, Alicante
  - LEO Pharma investigational site, Barcelona
  - LEO Pharma investigational site, Cadiz
  - LEO Pharma investigational site, Esplugues de Llobregat
  - LEO Pharma investigational site, Fuenlabrada
  - LEO Pharma investigational site, Granada
- United Kingdom (5):
  - LEO Pharma investigational site, Ipswich
  - LEO Pharma investigational site, Kings Lynn
  - LEO Pharma investigational site, Lincoln
  - LEO Pharma investigational site, London
  - LEO Pharma investigational site, Walsall

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at sites in 7 countries (Australia, Belgium, Canada, Spain, France, United Kingdom, and Poland).
Pre-assignment Details: Participants were randomized 3:1 to treatment with delgocitinib cream 20 mg/g or cream vehicle.
Groups:
- Delgocitinib Cream: Participants were randomized to twice-daily topical applications of delgocitinib cream 20 mg/g for a 16-week treatment period followed by a follow-up period of 2 weeks for assessment of safety.
  Delgocitinib cream: Cream for topical application.
- Cream Vehicle: Participants were randomized to twice-daily applications of cream vehicle for a 16-week treatment period followed by a follow-up period of 2 weeks for assessment of safety.
  Cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active medical ingredient.
Period: Overall Study
Arm/Group | Delgocitinib Cream | Cream Vehicle
Started | 74 | 24
Completed | 71 | 21
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delgocitinib Cream | Cream Vehicle | Total
Number analyzed (Participants) | 74 | 24 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 24 | 98
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.7) | 14.7 (1.6) | 14.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 12 | 58
  Male | 28 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 8
  Not Hispanic or Latino | 62 | 21 | 83
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 69 | 20 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 1 | 7
  Belgium | 2 | 0 | 2
  Poland | 23 | 9 | 32
  United Kingdom | 5 | 2 | 7
  Australia | 10 | 4 | 14
  France | 11 | 5 | 16
  Spain | 17 | 3 | 20
IGA-CHE score [Count of Participants; unit: Participants] — The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    Clear | 0 | 0 | 0
    Almost clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 56 | 18 | 74
    Severe | 18 | 6 | 24
HECSI score [Mean (Standard Deviation); unit: scores on a scale] — The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score), with a higher score indicating greater severity.
  scores on a scale | 70.9 (37.8) | 76.2 (39.7) | 72.2 (38.1)
HESD itch score (weekly average) [Mean (Standard Deviation); unit: scores on a scale] — The Hand Eczema Symptom Diary (HESD) itch score is one component of the HESD eDiary. In the HESD eDiary, participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. Population: Data is missing for 1 participant in the delgocitinib cream group.
  scores on a scale
    number analyzed (Participants) | 73 | 24 | 97
    (all) | 5.56 (2.59) | 5.91 (3.01) | 5.65 (2.69)
HESD pain score (weekly average) [Mean (Standard Deviation); unit: scores on a scale] — The Hand Eczema Symptom Diary (HESD) pain score is one component of the HESD eDiary. In the HESD eDiary, participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. Population: Data is missing for 1 participant in the delgocitinib cream group.
  scores on a scale
    number analyzed (Participants) | 73 | 24 | 97
    (all) | 5.20 (2.75) | 5.65 (3.49) | 5.31 (2.94)
HESD score (weekly average) [Mean (Standard Deviation); unit: scores on a scale] — The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. The HESD score is derived as the average of the 6 signs and symptoms. Population: Data is missing for 1 participant in the delgocitinib cream group.
  scores on a scale
    number analyzed (Participants) | 73 | 24 | 97
    (all) | 5.63 (2.26) | 5.75 (3.00) | 5.66 (2.45)
CDLQI score [Mean (Standard Deviation); unit: scores on a scale] — The Children's Dermatology Life Quality Index (CDLQI) is a validated questionnaire consisting of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week. Each question is scored from 0 (no impact) to 3 (high impact). The CDLQI score is the sum of the 10 items (score ranging from 0 to 30).
  scores on a scale | 8.5 (5.5) | 9.6 (6.8) | 8.8 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With IGA-CHE Treatment Success at Week 16
Description: The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is a 5 point scale used in clinical trials to rate the severity of the subject's CHE from 0 (clear) to 4 (severe). Treatment success means a score of 0 (clear) or 1 (almost clear) with a ≥2 step improvement from baseline.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
Participants | 47 | 7
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; Based on the primary estimand 'composite'. Data considered non-response after initiation of rescue treatment or after permanent discontinuation of IMP. Missing data imputed as non-response; Test type: Superiority; Bayesian — There are no p-values when performing a Bayesian analysis. Instead, the probability that the difference in the posterior distributions is > 0 is used; Historical information from LP0133-1401 (NCT04871711)/LP0133-1402 (NCT04872101) as prior information is used; Diff. in proportion of responders in % = 37.9 — There is no confidence interval when performing Bayesian analyses - instead a 95% credibility interval is used: 13.5% to 58.2%

2. Secondary Outcome: Number of Participants With HECSI-90 at Week 16
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score), with a higher score indicating greater severity. HECSI-90 is defined as at least 90% improvement in HECSI score from baseline.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
Participants | 53 | 9
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; Primary estimand: Composite. Data considered non-response after initiation of rescue treatment or after permanent discontinuation of IMP. Missing data imputed as non-response; Test type: Superiority; Bayesian — [p-value comment as in outcome 1, analysis 1]; Diff. in proportion of responders in % = 36.4 — There is no confidence interval when performing Bayesian analyses - instead a 95% credibility interval is used: 12.3% to 59.9%

3. Secondary Outcome: Number of Participants With Reduction of HESD Itch Score (Weekly Average) of ≥4 Points From Baseline at Week 16
Description: The Hand Eczema Symptom Diary© (HESD) is an instrument designed to assess severity of CHE signs and symptoms. The participants will assess the worst severity of 6 individual signs and symptoms of CHE from 0 (none) to 10 (severe) over the past 24 hours. The participants will complete the HESD on a daily basis in an eDiary.' This endpoint will only assess the 'itch' component for participants with a baseline HESD itch score (weekly average) of ≥4 points.
Time Frame: Week 16
Population: Data is not available for 20 participants in the Delgocitinib cream group and for 5 participants in the cream vehicle group.
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 54 | 19
Participants | 35 | 7
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; Test type: Superiority; Bayesian — [p-value comment as in outcome 1, analysis 1]; Diff. in proportion of responders in % = 31.7 — There is no confidence interval when performing Bayesian analyses - instead a 95% credibility interval is used: 5.6% to 51.1%

4. Secondary Outcome: Number of Participants With Reduction of HESD Pain Score (Weekly Average) of ≥4 Points From Baseline at Week 16
Description: The Hand Eczema Symptom Diary© (HESD) is an instrument designed to assess severity of CHE signs and symptoms. The participants will assess the worst severity of 6 individual signs and symptoms of CHE from 0 (none) to 10 (severe) over the past 24 hours. The participants will complete the HESD on a daily basis in an eDiary.' This endpoint will only assess the 'pain' component for participants with a baseline HESD pain score (weekly average) of ≥4 points.
Time Frame: Week 16
Population: Data is not available for 25 participants in the Delgocitinib cream group and for 9 participants in the cream vehicle group.
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 49 | 15
Participants | 31 | 5
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; Test type: Superiority; Bayesian — [p-value comment as in outcome 1, analysis 1]; Diff. in proportion of responders in % = 31.2 — There is no confidence interval when performing Bayesian analyses - instead a 95% credibility interval is used: 8.7% to 49.4%

5. Secondary Outcome: Number of Participants With Reduction of HESD Score (Weekly Average) of ≥4 Points From Baseline at Week 16
Description: The Hand Eczema Symptom Diary© (HESD) is an instrument designed to assess severity of CHE signs and symptoms. The participants will assess the worst severity of 6 individual signs and symptoms of CHE from 0 (none) to 10 (severe) over the past 24 hours. The participants will complete the HESD on a daily basis in an eDiary.' The final HESD score is an average of these 6 individual scores. This endpoint will only assess the score for participants with a baseline HESD itch score (weekly average) of ≥4 points.
Time Frame: Week 16
Population: Data is not available for 20 participants in the Delgocitinib cream group and for 8 participants in the cream vehicle group.
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 54 | 16
Participants | 30 | 5
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Bayesian — [p-value comment as in outcome 1, analysis 1]; Diff. in proportion of responders in % = 25.1 — There is no confidence interval when performing Bayesian analyses - instead a 95% credibility interval is used: 3.9% to 42.3%

6. Secondary Outcome: Number of Participants With IGA-CHE Treatment Success at Week 2
Description: as for outcome 1
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
Participants | 16 | 1
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; The primary estimand using the composite strategy is used for the analysis. Data is considered non response after initiation of rescue treatment or after permanent discontinuation of IMP. Missing data is imputed as non-response; Test type: Superiority; p = 0.0054, Regression, Logistic; Risk Difference (RD) = 17.47, 95% CI 2-sided [5.16 to 29.78] — Risk difference estimated using logistic regression stratified by baseline IGA-CHE score

7. Secondary Outcome: Number of Participants With IGA-CHE Treatment Success at Week 4
Description: The Investigator's Global Assessment for chronic hand eczema© (IGA-CHE) is a 5 point scale used in clinical trials to rate the severity of the subject's CHE from 0 (clear) to 4 (severe). Treatment success means a score of 0 (clear) or 1 (almost clear) with a ≥2 step improvement from baseline.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
Participants | 28 | 4
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0248, Regression, Logistic; Risk Difference (RD) = 21.21, 95% CI 2-sided [2.69 to 39.72] — Risk difference estimated using logistic regression stratified by baseline IGA-CHE score

8. Secondary Outcome: Number of Participants With IGA-CHE Treatment Success at Week 8
Description: as for outcome 7
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
Participants | 36 | 9
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3320, Regression, Logistic; Risk Difference (RD) = 11.08, 95% CI 2-sided [-11.30 to 33.46] — Risk difference estimated using logistic regression stratified by baseline IGA-CHE score

9. Secondary Outcome: Number of Participants With IGA-CHE Treatment Success at Week 12
Description: as for outcome 7
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
Participants | 43 | 6
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0016, Regression, Logistic; Risk Difference (RD) = 33.02, 95% CI 2-sided [12.51 to 53.52] — Risk difference estimated using logistic regression stratified by baseline IGA-CHE score

10. Secondary Outcome: Change in CDLQI Score From Baseline to Week 16
Description: The Children's Dermatology Life Quality Index (CDLQI) is a validated questionnaire consisting of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week. Each question is scored from 0 (no impact) to 3 (high impact). The CDLQI score is the sum of the 10 items (score ranging from 0 to 30); a high score is indicative of a poor quality of life.
Time Frame: Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
score on a scale | -5.57 (0.44) | -2.92 (0.78)
Statistical Analysis 1: Comparison: Delgocitinib Cream vs Cream Vehicle; Primary estimand: Composite. Data considered non-response by using WOCF (including the baseline value) after initiation of rescue treatment or after permanent discontinuation of IMP. Missing data imputed using WOCF (including the baseline value); Test type: Superiority; p = 0.0038, ANCOVA; Mean Difference (Net) = -2.65, 95% CI 2-sided [-4.42 to -0.88]

11. Secondary Outcome: Number of Treatment Emergent AEs From Baseline up to Week 18
Description: An adverse event (AE) will be considered treatment emergent if started after the first application of treatment, or started before the first application of treatment and worsened in severity after treatment.
Time Frame: Week 18
Measure: Number; unit: events
Arm/Group | Delgocitinib Cream | Cream Vehicle
Number analyzed (Participants) | 74 | 24
events | 77 | 19

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected during the 16 weeks of treatment + 2 weeks of follow-up.
Arm/Group | Delgocitinib Cream | Cream Vehicle
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/24
Other Adverse Events (participants affected / at risk) | 17/74 | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib Cream (N=74) | Cream Vehicle (N=24)
Nasopharyngitis (Infections and infestations) | 10 (12) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT05355818/Prot_SAP_000.pdf